CLINICAL TRIAL: NCT05526157
Title: FINErenone druG Utilization Study and Assessment of Temporal Changes Following Availability of Different Treatment Options in Patients With Chronic Kidney Disease and Type 2 Diabetes
Brief Title: An Observational Study, Called FINEGUST, to Learn More About How People With Chronic Kidney Disease and Type 2 Diabetes Are Treated and How the Introduction of New Treatment Options, Like Finerenone, Impacts Clinical Practice
Acronym: FINEGUST
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21956
Record Dates: First submitted 2022-08-19; First posted 2022-09-02 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes Mellitus
Keywords: Chronic kidney disease; Type 2 diabetes mellitus; Impaired kidney function; Non-steroidal mineralocorticoid receptor antagonist (nsMRA)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — finerenone; Sodium-Glucose Transporter 2 Inhibitors; Glucagon-Like Peptide-1 Receptor Agonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with CKD+T2D in Study period I: In the pre-finerenone approval period (Study period I), 4 new-user cohorts to be identified, based on the first use of any drug in these classes: SGLT2i, GLP-1 RA, sMRA, or nsMRA.
  Interventions: Drug: Sodium-glucose cotransporter 2 inhibitors (SGLT2i); Drug: Glucagon-like peptide-1 receptor agonists (GLP 1 RA); Drug: Steroidal mineral corticoid receptor antagonists (sMRA); Drug: Non-steroidal mineral corticoid receptor antagonists (nsMRA)
- Patients with CKD+T2D in Study period II: In the post-finerenone study period (study period II), 3 new-user cohorts will be identified: SGLT2i, GLP-1 RA, and finerenone.
  Interventions: Drug: Finerenone (Kerendia, BAY 948862); Drug: Sodium-glucose cotransporter 2 inhibitors (SGLT2i); Drug: Glucagon-like peptide-1 receptor agonists (GLP 1 RA)

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY 948862) — Retrospective analysis using secondary data collection from various sources
  Groups: Patients with CKD+T2D in Study period II
Drug: Sodium-glucose cotransporter 2 inhibitors (SGLT2i) — Retrospective analysis using secondary data collection from various sources
Drug: Glucagon-like peptide-1 receptor agonists (GLP 1 RA) — Retrospective analysis using secondary data collection from various sources
Drug: Steroidal mineral corticoid receptor antagonists (sMRA) — Retrospective analysis using secondary data collection from various sources
  Groups: Patients with CKD+T2D in Study period I
Drug: Non-steroidal mineral corticoid receptor antagonists (nsMRA) — Retrospective analysis using secondary data collection from various sources
  Groups: Patients with CKD+T2D in Study period I

SUMMARY:
This is an observational study in which data from people with chronic kidney disease (CKD) and type 2 diabetes (T2D) who have already started or will start CKD or T2D treatment are collected and studied. In observational studies, only observations are made without specified advice or interventions.

People receiving the following CKD or T2D treatments as recommended by their doctors will be included:

* Sodium-glucose cotransporter 2 inhibitors (SGLT2i),
* Glucagon-like peptide-1 receptor agonists (GLP-1 RA),
* Steroidal mineralocorticoid receptor antagonists (sMRA),
* Finerenone, a non-steroidal mineralocorticoid receptor antagonist (nsMRA)
* Other nsMRA (only in Japan)

Kidneys filter extra water and waste from the blood and make urine. CKD is a long-term, progressive decrease in the kidneys' ability to properly filter blood. In people with T2D, the body does not make enough of a hormone called insulin or does not use insulin well enough, resulting in high blood sugar levels that can cause damage to the kidneys. As a result, CKD can occur as a complication of T2D.

The new drug, finerenone, works by blocking certain proteins, called mineralocorticoid receptors. An increased stimulation of these proteins is thought to damage the kidneys. By lowering their stimulation, finerenone reduces the risk of progressive worsening of the kidney disease.

Finerenone is available and approved in several countries for doctors to prescribe to people with CKD and T2D.

The main purpose of the study is to collect and describe characteristics of participants in each treatment group who have started or will start treatment before and after finerenone became available.

To do this, the researchers will collect data on:

* Patient characteristics (e.g., age sex) of the participants
* Clinical characteristics (e.g., history of CKD and T2D, heart and liver health, other health problems) of the participants
* Treatments for T2D and CKD
* Other medications used

Data will be grouped by type of treatment that is initiated (e.g., SGLT2i, a GLP-1 RA, a sMRA, finerenone, or other nsMRA). Two time periods will be compared. Study period I is the time until finerenone became available in the respective country, starting from 2012 (2014 for Japan). Study period II will begin when finerenone becomes available in the respective country and will end at the end of the study (planned in September 2024).

Researchers will also collect data on treatment patterns and changes for each type of treatment in both time periods.

Health care data will be collected from various sources in five countries (e.g., Denmark, the Netherlands, Spain, Japan, and the US).

The patients will receive their treatment as prescribed by their doctors during routine practice according to the approved product information.

Each patient will be in the study from first use (in Study period I and II) of one of the listed drug classes until:

* End of study
* The data are somehow no longer available
* The patient leaves or has to leave the study

ELIGIBILITY:
Inclusion Criteria:

* Active registration or continuous enrolment for at least 12 months in 1 of the selected data sources before the index date
* No recorded prescription or dispensing of any medication in the class during the 12 months before the index date
* Age 18 years or older as of the index date
* Diagnosis of T2D on or before the index date
* Diagnosis of CKD on or before the index date

Exclusion Criteria:

* Type 1 diabetes identified by appropriate algorithms in each participating data source
* Kidney cancer on or before the index date
* Kidney failure

  -- Maintenance dialysis on or before the index date
* Kidney transplantation on or before the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted using data from data sources in 5 countries: Denmark (the Danish National Health Registers), Japan (the Japan Chronic Kidney Disease Database), the Netherlands (PHARMO), Spain (the Valencia Health System Integrated Database), and the US (Optum). For each database, the source population will include patients who fulfil an electronic algorithm for CKD and T2D.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Descriptive summary of baseline patient characteristics | Baseline study periods I and II
  Demographic (Age, Sex, Race and Socioeconomic status ) and clinical characteristics (markers of severity of T2D and of kidney dysfunction ) data will be collected.
Descriptive summary of patient comorbidities | Baseline study periods I and II
  History of coronary heart disease, cerebrovascular disease, peripheral vascular disease, hypertension, hypercholesterolemia, Congestive heart failure, Severe liver disease, Other comorbidities measured by the Charlson or similar comorbidity indices. Lifestyle factors as Body mass index (BMI) or evidence of obesity, Smoking status, and alcohol abuse and alcohol abuse-related conditions, as available in each data source.
Descriptive summary of patient comedications | Baseline study periods I and II
  Medications for T2D, CKD and other relevant medications.

SECONDARY OUTCOMES:
Descriptive summary of changes over time in treatments in the new-user cohorts | From Day 1 until Censor Day (at the earliest of death, disenrolment, exclusion criteria during follow-up, or end of the study period) [up to 114 months for study period I and up to 39 months for study period II].
Descriptive summary of temporal changes in the baseline characteristics of medication-specific cohorts | Baseline up to 114 months for study period I and up to 39 months for study period II

CONTACTS AND LOCATIONS:
Locations (5):
- Optum CDM, Eden Prairie, Minnesota, United States
- Many Locations, Multiple Locations, Denmark
- Many Locations, Multiple Locations, Japan
- Many Locations, Multiple Locations, Netherlands
- Many Locations, Multiple Locations, Spain

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Johannes CB, Coleman CI, Kovesdy CP, Khan AM, Ziemiecki R, Layton JB, Vizcaya D, Liu F, Oberprieler NG. Temporal Changes in SGLT2 Inhibitor and GLP-1 Receptor Agonist Use in Patients with Chronic Kidney Disease and Type 2 Diabetes, 2012-2023: A US Cohort Study. Diabetes Ther. 2025 Dec 9. doi: 10.1007/s13300-025-01825-5. Online ahead of print. PMID 41364416